CLINICAL TRIAL: NCT02251197
Title: A Randomised, Double-blind, Placebo-controlled, Clinical Trial to Evaluate the Safety and Tolerability in 108 Patients (18 Per Dose Group) With Acute Ischemic Stroke After Intravenous Administration From 6 to 72 Hours of BIII 890, as Loading Dose Followed by Maintenance Dose, in Escalating Dose Panels From 87.5 mg up to 1495 mg (Total Dose)
Brief Title: Safety and Tolerability of BIII 890 in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 599.3
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — BIII 890 CL

ARMS (2):
- BIII 890 CL (Experimental): escalating doses
  Interventions: Drug: BIII 890 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIII 890 CL
  Arms: BIII 890 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety, tolerability and pharmacokinetic characteristics of BIII 890 after intravenous infusion in acute ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or above
* Patients with an acute onset of a focal neurological deficit secondary to a lesion presumed to be ischemic in etiology involving the carotid and/or vertebrobasilar artery territories
* Onset of symptoms within 24 hours prior to initiation of administration of study drug. If the patient has awakened from sleep with the deficit, the time of onset will be considered as the last time he/she was normal
* Stroke symptoms are to be present for at least 1 hour and are still present at randomisation. Symptoms must be distinguishable from an episode of generalised ischemia (i.e. syncope), seizure, migraine or hypoglycaemic disorder
* Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each Patient (or the subject's representative or relatives, depending on local regulations) according to Good Clinical Practice and regulatory and legal requirements of the participating country. Patients who are unable to sign but who are able to understand the meaning of participation in the study may give an oral witnessed informed consent. These patients have to make clear undoubtfully that they are wiling to participate voluntarily and must be able to understand an Explanation of the contents of the Information sheet
* Patient's life expectancy is at least 30 days (investigator's judgement)

Exclusion Criteria:

* Presence of only minor stroke symptoms as characterised by a NIH score of < 4 at the time of randomisation
* Severe obtundation as defined by a NIH Stroke Scale score of ≥ 2 using the Level of Consciousness category; including coma or severe stupor
* Any patient with a concurrent, severe neurological disease

  * Dementia, multi-infarct dementia
  * Multiple sclerosis
  * Previous stroke with residual deficit (i.e. pre-stroke modified Rankin Scale (mRS) must be ≤ 1). Tomographic or clinical evidence of brain stem infarct, any intracranial haemorrhage, primary or metastatic brain tumour, meningioma, or other space occupying lesion (e.g., subdural or epidural haematoma)
  * Patient with history of seizure related or not to their stroke diagnosis, except seizure secondary to fever in the childhood
* Any patients with a concurrent mental deficit (e.g., AXIS-I psychiatric disorders as defined by the Diagnostic and Statistical Manual (DSM) IV criteria: schizophrenia, mood disorders (mania or major depression), psychotic/delusional disorders, a recent history (6 months) or current evidence of alcohol or recreational drug abuse
* Baseline blood glucose values below 2.75 mmol/l (hypoglycaemia) or above 22.0 mmol/l (hyperglycaemia)
* Sustained supine hypertension during the baseline period, and prior to randomisation, as defined as two readings 30 minutes apart with a systolic blood pressure ≥ 220 mmHg and/or a diastolic blood pressure ≥ 120 mmHg; and/or clinical diagnosis of malignant hypertensive crisis accompanied by other signs or symptoms (e.g. nausea, vomiting, obtundation, etc.) or complications (e.g. papilledema, retinal haemorrhage, hematuria, or congestive heart failure)
* Patients with known history of orthostatic hypotension, fainting spells or blackouts. Hypotension as defined by a systolic blood pressure ≤ 90 mmHg or a diastolic blood pressure ≤ 50 mmHg
* Patients currently on oral anticoagulants. A time window of at least two days should be observed when such a treatment has been administered and stopped before the beginning of the trial
* Known history of a serious, advanced, unstable or terminal illness that in the opinion of the clinical investigator may interfere with the trial by confounding the results or pose an additional risk:

  * cardiogenic shock, congestive heart failure (NYHA Class III-IV), acute myocardial infarction or history of a myocardial infarction within the past three months, unstable angina
  * renal failure, severe hepatic disease, unstable gastrointestinal, pulmonary, metabolic, immunological, hormonal disorders
  * cancer (except local skin cancers, e.g.: basal or squamous carcinoma)
  * HIV+
* Females who are lactating or pregnant (as determined by a pregnancy test during screening) or of childbearing potential
* Current or recent (within 3 months) participation in another investigational drug protocol
* Patient cannot be followed for 30 days (according to the judgement of the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2001-07; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 45 days
Number of patients with clinically relevant findings in vital signs | up to 30 days
Number of patients with clinically relevant findings in electrocardiogram (ECG) | up to 45 days
Number of patients with clinically relevant findings in laboratory evaluation | up to 45 days

SECONDARY OUTCOMES:
Maximum concentration in plasma | up to 120 hours after drug administration
Time to reach maximum concentration in plasma | up to 120 hours after drug administration
Terminal elimination half-life | up to 120 hours after drug administration
Terminal rate constant | up to 120 hours after drug administration
Area under the plasma concentration-time curve | up to 120 hours after drug administration
Mean residence time | up to 120 hours after drug administration
Plasma clearance | up to 120 hours after drug administration
Volume of distribution at steady state | up to 120 hours after drug administration
Glutamate plasma concentrations | up to 72 hours after start of infusion
Change in modified Rankin Scale | Baseline, day 30
Barthel Index | Day 30
Change in NIH stroke scale | Baseline, day 1, 3, 7 and 30